CLINICAL TRIAL: NCT02327130
Title: Changes in Exhaled 13CO2/12CO2 Breath Delta Value as an Early Indicator of Infection in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isomark, LLC (Industry)
Collaborators: University of Florida (Other); Ohio State University (Other); Washington University School of Medicine (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Canary01; NCT02258022 (obsolete NCT alias)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exhaled Breath (Experimental): Exhaled breath samples will be collected 6 times per day and blood samples will be collected once per day for 7 days. Subjects will be followed for an additional 3 days. We will use the Isomark Canary™ to determine the BDV of breath samples collected during this study. Analysis results of these samples will be combined with data that is abstracted from the subjects' medical records.
  Interventions: Device: Isomark Canary™

INTERVENTIONS:
Device: Isomark Canary™ — Isomark, LLC is a Madison, Wisconsin-based company that has developed an investigational device, the Isomark Canary™, that is intended to determine the breath delta value of breath samples collected from critically ill patients.

SUMMARY:
Carbon-12 and carbon-13 are naturally-abundant isotopes in exhaled breath carbon dioxide. The ratio of carbon-13 to carbon-12 in exhaled breath is known as the breath delta value (BDV). This study is seeking to determine if the breath delta value of critically ill adults is an early indicator of the onset of infection that may lead to sepsis.

DETAILED DESCRIPTION:
Sepsis is a major complication for any patient, and its management is an acknowledged challenge for intensivists. Sepsis has unpredictable onset and progression, and is a leading cause of death in ICUs with a mortality rate of 30-50%. Annually in the US, 1.4M cases involve hospitalization, 750,000 cases of severe sepsis or septic shock, and ~260,000 cases of sepsis related death have been reported in recent years. Current experience of UF Health investigators in surgical ICUs is 1 -2 sepsis, severe sepsis, or septic shock patients per day, of which ~10% are trauma patients. Of trauma patients, ~8% develop sepsis during their ICU stay.

Breath delta value is hypothesized to be a biomarker of infection. Breath delta value is not a defined clinical outcome related to human health, because this study is seeking to establish breath delta value as a biomarker of infection. This study is measuring the feasibility of the Isomark Canary™ device. If the Canary does not detect a significant decrease in breath delta value in those subjects who subsequently get an infection, it will not be feasible to use it for this purpose.

Breath delta value will be collected to determine its relationship to infection, no health outcomes are being measured.

This study is designed to determine if the BDV of adult ICU patients is an early indicator of the onset of infection that may lead to sepsis.

The objectives of this study are: (1) to measure variation of BDV with time in adult ICU patients who agree to participate as research subjects; (2) to determine the magnitude of change of BDV in subjects who are subsequently diagnosed with severe infection and sepsis; (3) to define variation of BDV in adult trauma subjects who do not develop severe infection.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. critically ill patient admitted to trauma or surgical ICU
3. expected duration of hospital stay at least 120 hours (five days) from time of study enrollment
4. subject/LAR speaks a language of which the IRB has approved a consent form

Exclusion Criteria:

1. known infection at the time of enrollment per infection definitions in section 6.2
2. known use of systemic antibiotic, antimicrobial and/or antifungal therapy within the last 7 days (See Antibiotic Use section below)
3. prolonged antibiotic or antimicrobial use during the perioperative period (See Antibiotic Use section below)
4. currently active cancer, or receiving treatment for cancer (including but not limited to: radiation, chemotherapy, systemic orals, etc)
5. receiving high frequency ventilatory support
6. if not intubated, unable to cooperate with providing a breath sample
7. expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family/medical team (e.g., likely to withdraw life support measures within 24 hrs of screening)
8. female who is pregnant or lactating (negative serum or urine pregnancy test results within 48 hours of enrollment or to be performed during screening)
9. prisoner
10. known participation in an interventional research study within 30 days prior to enrollment (note: to be eligible, any interventional treatment must have ended at least 30 days ago)
11. Individuals who are directly affiliated with sponsor or study staff, or their immediate families. Immediate family is defined as spouse, domestic partner, parent, child, or sibling whether legally adopted or biological.
12. Any patient that is deemed unfit for study participation, per the Investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Florida Health, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Isomark, LLC, Madison, Wisconsin

REFERENCES:
- [Derived] O'Rourke AP, Buckman SA, Evans DC, Kerwin AJ, Breunig EA, Butz DE. Changes in exhaled 13CO2/12CO2 breath delta value as an early indicator of infection in intensive care unit patients. J Trauma Acute Care Surg. 2019 Jan;86(1):71-78. doi: 10.1097/TA.0000000000002097. PMID 30575683

RESULTS

PARTICIPANT FLOW:
Groups:
- Isomark Canary: All subjects were enrolled were at risk for developing infections during the study but did not currently exhibit signs of ongoing infection. The 'at risk' enrolled subjects utilized the Isomark Canary to take exhaled breath samples to assess for infection status.
Period: Overall Study
Arm/Group | Isomark Canary
Started | 32
Completed | 20
Not Completed | 12
Not completed — Discharged in less than 5 days | 5
Not completed — Physician Decision | 2
Not completed — Unable to provide breath sample | 1
Not completed — Incorrectly place ventilator adaptor | 1
Not completed — Met exclusion criteria | 3

BASELINE CHARACTERISTICS:
Groups:
- Critically Ill Subjects at Risk for Infection: Critically ill adult ICU subjects who are not suspected of having an infection at the time of ICU admission were enrolled as study subjects.
Arm/Group | Critically Ill Subjects at Risk for Infection
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Breath Delta Value
Description: The variation in breath delta value was assessed regardless of infection status. Exhaled breath samples were collected from participants upon enrollment and every four hours thereafter until the end of the subject's study duration per protocol. Each subject was used as its own control for the purpose of trend analysis.The first breath sample collected was considered an individual's "baseline" sample. The change in the breath delta value was calculated from this baseline sample.
Time Frame: Baseline to ICU discharge or 7 days, whichever came first
Measure: Mean (Standard Error); unit: parts per mil (‰)
Groups:
- Exhaled Breath: Exhaled breath samples were collected 6 times per day for 7 days. We will use the Isomark Canary™ to determine the BDV of breath samples collected during this study.
Arm/Group | Exhaled Breath
Number analyzed (Participants) | 20
parts per mil (‰) | 0.44 (1.09)

2. Secondary Outcome: Number of Participants With an Infection Diagnosis
Description: Daily analysis infection status from blood samples given from each participant.
Time Frame: Days 1 through 7
Measure: Number; unit: Participants
Groups:
- Infection Diagnosis: An endpoint adjudication committee (EAC), composed of three independent senior infectious disease experts, not involved in the subject clinical care, reviewed each study subjects' data to determine the clinical time and date of infection. Each EAC member independently reviewed the subject cases and completed the EAC Infection Status case report form. In cases where an infection developed the EAC placed a time and date stamp for time of first suspicion of infection and confirmation based on clinical judgement culture, or diagnostic imaging.
Arm/Group | Infection Diagnosis
Number analyzed (Participants) | 20
Participants | 11

3. Other Pre Specified Outcome: Positive and Negative Predictive Value of BDV for Infection Diagnosis
Description: Based on an ROC analysis the optimal cutoff value for indicating the presence of infection using the BDV is 1.4‰.
  Based on this cutoff value the sensitivity and specificity were calculated. Sensitivity, or the true positive rate, is the proportion of actual positives that are correctly identified. In this case, the sensitivity is the percentage of people who have an infection and were identified by the Isomark Canary as having an 'infection'.
  The specificity, or the true negative rate, is the promotion of actual negatives that are correctly identified as negative. In this case, the specificity is the proportion of people without infections that were correctly classified by the Isomark Canary as having 'no infection'.
Time Frame: 7 days
Measure: Number; unit: percent
Groups:
- Sensitivity: Percent sensitivity for BDV to predict an infection
- Specificity: Percent specificity for BDV to predict an infection
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 20 | 20
percent | 90.1 | 66.7

ADVERSE EVENTS:
Time Frame: 10 days per subject, throughout enrollment period April 2015 to December 2017.
Groups:
- At Risk for Infection: All subjects were enrolled were at risk for developing infections during the study but did not currently exhibit signs of ongoing infection.
Arm/Group | At Risk for Infection
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02327130/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02327130/SAP_001.pdf